CLINICAL TRIAL: NCT02339038
Title: A Phase IV Pilot Study to Assess Community-Based Treatment Efficacy in Chronic Hepatitis C Monoinfection and Coinfection With HIV in the District of Columbia
Brief Title: Community-based Treatment of Chronic Hepatitis C Monoinfection and Coinfection With HIV in the District of Columbia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15N064; 15-CC-N064 (Other: NIH); 999915064 (Other: NIHCC)
Record Dates: First submitted 2015-01-14; First posted 2015-01-15 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2017-06

CONDITIONS: HCV HIV
Keywords: Community Based Research; Hepatitis C Virus and Human Immunodeficiency Virus; Ledipasvir/Sofosbuvir; Fixed Dose Combination; Sustained Viral Response
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome | interventions — ledipasvir; Sofosbuvir; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Standard of Care (Other): Standard of care treatment using Ledipasvir 90 mg and Sofosbuvir 400 mg fixed dose combination by mouth daily for 2, 3, or 6 months
  Interventions: Drug: Ledipasvir 90 mg and Sofosbuvir 400 mg

INTERVENTIONS:
Drug: Ledipasvir 90 mg and Sofosbuvir 400 mg — Ledipasvir 90 mg and Sofosbuvir 400 mg fixed dose combination as per standard of care treatment guidelines
  Other Names: Harvoni

SUMMARY:
Background:

- Treatment for Hepatitis C has changed a lot in the past 2 years. Most of this change comes from a combination of medicines that is yielding high cure rates. But its long-term effects are uncertain. One problem is that a lot of people need the treatment, but only a few specialists can give it. The success rate for Hepatitis C treatment by primary care doctors, nurse practitioners, or physician assistants is largely unknown. Researchers want to see how provider type affects treatment outcomes. They will conduct a large, community-based study in the District of Columbia.

Objectives:

- To see if people can be treated for Hepatitis C safely and successfully in community-based health centers.

Eligibility:

- Adults who need treatment for chronic Hepatitis C infection.

Design:

* Participants will be screened with blood tests. Their current medicines will be reviewed.
* Participants will give researchers access to their medical records. Researchers will follow participants through these records.
* Participants will see a primary care or infectious disease provider. The provider will tell them about their treatment. They will be told how often they will visit the provider and how often they will have their blood drawn. They will get a calendar of study visits.
* Participants will take Harvoni for 8, 12, or 24 weeks. They will visit their care provider monthly.
* Participants will have monthly follow-up visits for up to 3 months after they finish their medicine.
* Participants will have yearly follow-up visits with their care provider for up to 10 years.

DETAILED DESCRIPTION:
Treatment for hepatitis C has been revolutionized in the last 2 years with the advent of combination antiviral therapy yielding high cure rates; although, the long term effects of treatment remain uncertain. Use of these medications has been limited to clinical trial settings typically by highly specialized care teams in tertiary care hospitals. As the prevalence of hepatitis C is significant, there exists a significant imbalance between patients who require treatment and specialists who provide treatment. Success rates in treatment of hepatitis C by primary care doctors or physician extenders, such as nurse practitioners or physician assistants, is largely unknown.

As such, we propose the first community-based, large scale, longitudinal study of directly acting antiviral (DAA)-based treatment for chronic hepatitis C, set in the District of Columbia. Within this study, approximately 600 HCV genotype 1 monoinfected and HCV/HIV coinfected subjects will be treated with ledipasvir/sofosbuvir (90 mg/400 mg) fixed dosed combination for 8-24 weeks, based on the medication labeling instructions, and followed for both immediate (SVR12) and long term (comorbid disease, cirrhosis, hepatocellular carcinoma, transplantation and mortality) outcomes over a 10 year study period. The study will be conducted exclusively in the District of Columbia clinics associated with the NIH DC Partnership for AIDS/HIV Progress (DC PFAP), which serves a population comprised primarily of minorities, with a high degree of negative predictors of treatment response. In this study, participants will be assigned to treatment either by (1) an ID or hepatology specialist, (2) primary care provider, or (3) physician extender. Please see Figure 1 study schema for an approximate distribution of subjects. Each of these provider groups will undergo uniform training on treatment of hepatitis C and management of adverse events prior to initiation of study. All subjects will sign informed consent and agree to treatment and follow up phases of the study. During the course of the study, subjcts will be clinically evaluated based on American Association for the Study of Liver Diseases (AASLD)/ the Infectious Diseases Society of America (IDSA) guidelines for the management of hepatitis C. Clinical data from subjects will be captured in a city wide cohort database, which will store guideline-driven data points from each clinic visit within the network.

Through this trial we will explore the efficacy of managing hepatitis C subjects with directly acting antiviral therapy in an urban, community-based setting, and investigate the effect of provider type (specialist, primary care, or physician extender) on treatment outcome. We will detail the safety and tolerability of this treatment. We will assess variability in treatment outcomes between monoinfected and HIV-coinfected subjects. Finally, we will evaluate the public health impact of large-scale treatment of HCV infected subjects in preventing long-term clinical outcomes. As the first interferon (IFN)- and ribavirin (RBV)-free, urban community-based treatment utilizing new standard of care criteria, this study will serve as a model for implementation of similar practice patterns globally.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male or female at least 18 years of age at time of screening who is determined to be eligible based on evaluation by a treating provider,
  2. Documentation of genotype 1 (GT-1) infection, liver fibrosis staging by any AASLD/IDSA guideline approved measurement, and HIV status determination.
  3. Chronic HCV genotype-1 infection prior to study enrollment. Chronic HCV-infection is defined as the following: positive for anti-HCV Ab or HCV RNA at least 6 months before screening, and positive for HCV RNA and anti-HCV Ab at the time of screening
  4. Compensated liver disease, both with and without cirrhosis, as determined clinically by referring provider
  5. If coinfected with HIV, stable HIV disease as determined by a treating provider
  6. Subjects must be able to understand and adhere to the study visit schedule and all other protocol requirements, and must voluntarily sign and date an informed consent form, approved by an Institutional Review Board (IRB), prior to the initiation of any screening or study specific procedures.

EXCLUSION CRITERIA:

1. Women who are pregnant or breastfeeding
2. Screening laboratory analyses showing any of the following abnormal laboratory results:

   - Estimated Glomerular Filtration Rate (eGFR) < 30 mL/min as estimated by the Modification of Diet in Renal Disease (MDRD) equation (utilized by LabCorp):

   eGFR = 175 times SerumCr(-1.154) age(-0.203 1.212 (if patient is black) 0.742 (if female)
3. Diagnosis of hepatocellular carcinoma as defined by pre-screening medical history
4. Any other conditions in the opinion of the investigator that would interfere with the compliance or endpoints of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2015-01-07; Primary Completion 2016-06-15 (Actual); Study Completion 2018-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Masur, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (2):
- United States (2):
  - Unity Health Care, Inc./DC General, Washington D.C., District of Columbia
  - Family Medical and Conseling Services, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohd Hanafiah K, Groeger J, Flaxman AD, Wiersma ST. Global epidemiology of hepatitis C virus infection: new estimates of age-specific antibody to HCV seroprevalence. Hepatology. 2013 Apr;57(4):1333-42. doi: 10.1002/hep.26141. Epub 2013 Feb 4. PMID 23172780
- [Background] Denniston MM, Jiles RB, Drobeniuc J, Klevens RM, Ward JW, McQuillan GM, Holmberg SD. Chronic hepatitis C virus infection in the United States, National Health and Nutrition Examination Survey 2003 to 2010. Ann Intern Med. 2014 Mar 4;160(5):293-300. doi: 10.7326/M13-1133. PMID 24737271
- [Background] Branch AD, Van Natta ML, Vachon ML, Dieterich DT, Meinert CL, Jabs DA; Studies of the Ocular Complications of AIDS Research Group. Mortality in hepatitis C virus-infected patients with a diagnosis of AIDS in the era of combination antiretroviral therapy. Clin Infect Dis. 2012 Jul;55(1):137-44. doi: 10.1093/cid/cis404. Epub 2012 Apr 24. PMID 22534149
- [Derived] Kattakuzhy S, Gross C, Emmanuel B, Teferi G, Jenkins V, Silk R, Akoth E, Thomas A, Ahmed C, Espinosa M, Price A, Rosenthal E, Tang L, Wilson E, Bentzen S, Masur H, Kottilil S; ASCEND Providers. Expansion of Treatment for Hepatitis C Virus Infection by Task Shifting to Community-Based Nonspecialist Providers: A Nonrandomized Clinical Trial. Ann Intern Med. 2017 Sep 5;167(5):311-318. doi: 10.7326/M17-0118. Epub 2017 Aug 8. PMID 28785771

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Standard of care treatment using ledipasvir 90mg-sofosbuvir 400mg by mouth daily for 2, 3, or 6 months
Period: Overall Study
Arm/Group | Standard of Care
Started | 600
Completed | 0
Not Completed | 600

BASELINE CHARACTERISTICS:
Arm/Group | Standard of Care
Number analyzed (Participants) | 600
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 522
  >=65 years | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184
  Male | 416
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 589
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 578
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Achieve Sustained Viral Response (SVR12) 12 Weeks After the Stop of Treatment Drugs
Description: The primary outcome was the number of patients with sustained viral response measured 12 weeks after the stop of treatment. The viral response was assessed by serum HCV RNA concentrations lower than the limit of quantification (<15IU/mL).
Time Frame: At least 12 weeks after completion of medication
Population: The analyses included all patients who received at least one dose of ledipasvir-sofosbuvir
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care
Number analyzed (Participants) | 600
Participants | 516

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Standard of Care
All-Cause Mortality (participants affected / at risk) | 8/600
Serious Adverse Events (participants affected / at risk) | 0/600
Other Adverse Events (participants affected / at risk) | 76/600
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=600)
Fatigue (General disorders) | 45
Headache (Nervous system disorders) | 40

LIMITATIONS AND CAVEATS:
Although primary outcome is complete, the study remains active for prolonged observation and numerous secondary outcomes, with a projected closure date in 2025.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes